CLINICAL TRIAL: NCT01381653
Title: An Innovative HIV Prevention Intervention Using Social Networking Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Responsible Party: Principal Investigator, Jeffrey T. Parsons, Professor, Hunter College of City University of New York
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R03DA031607 (NIH)
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Sexual Risk; Substance Use
Keywords: sexual risk; substance use; HIV prevention; intervention acceptability and feasibility; young men who have sex with men
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Motivational Interviewing (Experimental): Eight 30-minute sessions utilizing Motivational Interviewing will be delivered to reduce substance use and sexual risk in a group of high risk young men who have sex with men.
  Interventions: Other: Behavioral: HIV prevention intervention

INTERVENTIONS:
Other: Behavioral: HIV prevention intervention — Substance using HIV-negative young men who have sex with men who engage in sexual risk and use social networking (Facebook) will be recruited and enrolled in a brief intervention utilizing Motivational Interviewing over chat window to reduce their substance use and sexual risk. They will also evaluate their intervention experience at the end of their eight sessions and post-assessment.
  Other Names: Reductions in sexual risk and substance use

SUMMARY:
An existing face-to-face HIV prevention intervention (The Young Men's Health Project, YMHP; R01DA20366) will be iteratively adapted and pilot-tested to target difficult to engage high-risk young men who have sex with men (YMSM) via online social networking and aims to reduce both high-risk sexual behavior and drug use.

DETAILED DESCRIPTION:
This pilot study entails a two-phase process. During Phase I, 15 former YMHP participants (intervention decliners and those who only completed one session) will participate in focus groups to advise us on the feasibility and pragmatic specifications of an HIV prevention intervention received via the IM (instant messaging) function of Facebook. Focus group transcripts will be examined to isolate key recommendations for modifying the intervention's structure and procedures. Focus groups will be reconvened for additional feedback on the modified intervention, followed by further adjustment. During Phase II, 40 high-risk YMSM (ages 18-29 and Facebook users) will be enrolled in a pilot of the modified intervention. The intervention will span 4 weeks and contain 8 bi-weekly 30 minute Motivational Interviewing (MI) chat-window sessions consisting of a sequential progression of intervention approaches tailored to each participant's readiness to change their drug use and high risk sexual behavior. Data from Phase II will include pre-post intervention behavioral risk assessments, as well as individual interviews with all 40 intervention participants for a qualitative evaluation regarding the feasibility and acceptability of the intervention's structure, and process. Findings from these interviews (and counselor focus group) will inform the fine-tuning of the intervention in preparation for a subsequent randomized control trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

Phase I:

For the focus group portion of the study (N=20), we will invite former YMHP participants who declined the intervention or only completed one session, agreed to be contacted for future studies, indicated using Facebook, are still between the ages of 18-29 and live in NYC.

Phase II:

To qualify for the intervention portion of the study, participants must report

1. at least 5 days of drug use (of 1 or more of the following drugs: cocaine, methamphetamine (MA), or ecstasy (MDMA) in the prior three months;
2. high-risk sexual behavior (1 or more acts of unprotected insertive or receptive anal sex with a male partner of unknown or HIV+ serostatus), in the prior three months;
3. biologically male;
4. age 18 to 29;
5. HIV-;
6. reliable Internet access;
7. Facebook use at least four times per week;
8. able to write in English given that intervention participation involves writing;
9. NYC residency.

Exclusion Criteria:

Participants will be excluded for any of the following reasons:

1. Unstable, serious psychiatric symptoms;
2. Currently suicidal/homicidal;
3. Evidence of gross cognitive impairment;
4. Self-reported current enrollment in a drug or HIV-related intervention or research study.

We exclude those with serious cognitive or psychiatric impairments because this would compromise ability to participate, regardless of whether these impairments are attributed to drug use. Such impairments would make completion of assessments difficult.

Excluded participants will be referred to local community health and social services resources, for which we have established linkages to facilitate access to care regardless of ability to pay.

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
feasibility and acceptability of intervention delivery | 1 month
  Participants (N=40) who received eight 30-minute sessions of Motivational Interviewing (to reduce substance use and sexual risk) over instant messaging on Facebook will be interviewed to evaluate the intervention delivery and structure, including their perceived connection with the counselor and concerns with receiving an intervention online.

CONTACTS AND LOCATIONS:
Overall Officials: Corina T Lelutiu-Weinberger, PhD, Principal Investigator — Hunter College, CUNY, Center for HIV/AIDS Educational Studies and Training
Locations (1):
- Hunter College, CUNY, Center for HIV/AIDS Educational Studies and Training, New York, New York, United States